CLINICAL TRIAL: NCT01824381
Title: Use of the Amniotic Membrane in Large Wound Epithelialization. Phase I Clinical Trial.
Brief Title: Use of the Amniotic Membrane in Large Wound Epithelialization
Acronym: MA/GH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Public Health Service, Murcia (Other); Universidad de Murcia (Other); Hospital Universitario Virgen de la Arrixaca (Other); MurciaSalud (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA/GH; 2011-004395-11 (EudraCT Number)
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Wounds
Keywords: extensive wounds; amniotic membrane; healing; patients; phase granulation
MeSH Terms: conditions — Wounds and Injuries | interventions — Biological Dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amniotic membrane in large wounds (Experimental)
  Interventions: Procedure: Place amniotic membrane in large wounds; Procedure: Obtaining and Cryopreservation of amniotic membrane; Drug: amniotic membrane

INTERVENTIONS:
Procedure: Place amniotic membrane in large wounds — After the process of obtaining the amniotic membrane, it must be processed, frozen and thawed.
  The wound is washed with saline and, if necessary it will be debrided. We will take microbiological control cultures. Then apply the amniotic membrane fragments sufficient to cover the wound by contacting the basal membrane of the amniotic membrane with granulation tissue.
  We will place a new membrane weekly to a maximum of 6 times.
Procedure: Obtaining and Cryopreservation of amniotic membrane
Drug: amniotic membrane

SUMMARY:
The purpose of this study is to analyze the security application of the amniotic membrane in extensive wounds in the granulation phase.

ELIGIBILITY:
Inclusion Criteria:

* Acute wounds in granulation phase with a minimum area of 100 cm2.
* Patients 18 or more years.
* Patients offering sufficient guarantees of adherence to protocol.
* Sign the written informed consent.
* Meet all inclusion criteria.

Exclusion Criteria:

* Patients with symptomatic chronic arterial insufficiency.
* Patients who are pregnant
* Patients in active lactation
* Patients physically fertile, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle or sexual orientation precludes intercourse with a man and women whose partners have been sterilized by vasectomy or other methods, UNLESS they are using reliable contraception. This method of contraception can be:

  * Complete abstinence from sexual intercourse
  * Surgical sterilization (tubal ligation)
  * Surgical sterilization of the partner (vasectomy)
  * Implanted or injectable hormonal contraceptives, oral *
  * Because hormonal contraceptives have a risk of thrombosis, should consider other methods of birth control.

These reliable contraception must be maintained during their participation in the study.

* Patients with heart, kidney, liver, systemic immune may influence the survival of the patient during the test.
* Participation in other clinical trials.
* Inability to understand informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety | Last revision at 3 years after surgery.
  No serious adverse events possibly, probably or definitely related with the procedure.
  No appearance of clinical inflammatory changes.

SECONDARY OUTCOMES:
Measurement of the wound area | 3 years
  To assess the effects of the application of the amniotic membrane on reepithelialization of wounds by measuring the wound area.
Evolution of local pain measured with a visual analog scale | 1 year
  To assess the effects of the application of amniotic membrane in the symptomatology of patients through the development of local pain measured with a visual analog scale.
Changes in the signaling pathways of TGFb. | 1 year
  To study the changes in the signaling pathways of TGFb in patients epithelium induced amniotic membrane.

CONTACTS AND LOCATIONS:
Overall Officials: Gregorio Castellanos-Escrig, MD, Principal Investigator — Clinical Universitary Hospital Virgen de la Arrixaca
Locations (1):
- Clinical Universitary Hospital Virgen de la Arrixaca, El Palmar, Murcia, Spain

REFERENCES:
- See also: Official web of Spanish Stem Cell Network — http://www.red-tercel.com
- See also: Fundación para la Formación e Investigación Sanitarias Región de Murcia — http://www.ffis.es
- See also: Official web of Health Service of Murcia Region. — http://www.murciasalud.es